CLINICAL TRIAL: NCT00719381
Title: Effect of Pioglitazone on Sputum Biomarkers of Inflammation and Lung Epithelial Repair in Cystic Fibrosis
Brief Title: Effect of Pioglitazone on Inflammation in Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paul Beringer (Other)
Responsible Party: Sponsor-Investigator, Paul Beringer, Associate Professor, University of Southern California
Organization: University of Southern California (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-07-00308; IND #: 101989
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Treatment of pioglitazone will consist of 15 mg once daily for 28 days followed by 30 mg once daily for 28 days (N=12)
  Interventions: Drug: Pioglitazone
- 2 (No Intervention): Patients in this arm will receive no intervention

INTERVENTIONS:
Drug: Pioglitazone — Treatment of pioglitazone will consist of 15 mg once daily for 28 days followed by 30 mg once daily for 28 days (N=12)
  Other Names: Actos
  Arms: 1

SUMMARY:
The purpose of this study is to determine the effect of pioglitazone on reducing airway inflammation in cystic fibrosis and characterize the amount and timecourse of pioglitazone elimination from the body.

DETAILED DESCRIPTION:
Progressive loss of lung function due to chronic infection and inflammation is the primary cause of morbidity and mortality in patients with CF. Current therapies directed at treatment of chronic P. aeruginosa infection (e.g. aerosolized tobramycin, azithromycin) provide short-term improvement in pulmonary function; however, persistence of the infection/inflammation causes the inevitable loss of lung function. PPARgamma is a nuclear transcription factor which is known to reduce activation of NFKB, a central mediator of airway inflammation in CF. Recent studies demonstrate that PPARgamma expression is reduced in patients with CF and may offer a potential therapeutic target to combat airway inflammation in CF. Pioglitazone is a thiazolidinedione whose principal pharmacological target it PPARgamma. The purpose of this pilot study is to determine the pharmacokinetics/pharmacodynamics of pioglitazone and effect on reducing airway inflammation in cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Clinically stable (FEV1 within 10% of baseline)
* FEV1 > 40% predicted

Exclusion Criteria:

* History of hypoglycemic events
* Hepatic disease (AST, ALT > 2.5x ULN)
* Renal disease (GFR < 60 ml/min - 1.73m2)
* Currently receiving beta-blocker, oral corticosteroids, statin, angiotensin receptor blocker, trimethoprim-sulfamethoxazole, gemfibrozil, or rifampin therapies.
* Allergy to thiazolidinediones
* Pregnancy or attempting to conceive, breast feeding
* Hematocrit < 30
* Congestive heart failure
* Pulmonary hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To determine the effect of pioglitazone on sputum biomarkers of lung inflammation and remodeling. | 83 days

SECONDARY OUTCOMES:
To characterize the pharmacokinetics, pharmacodynamics and safety of pioglitazone in patients with cystic fibrosis. | 83 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Beringer, Pharm.D., Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States